CLINICAL TRIAL: NCT03568864
Title: The Acute Effect of a High Nucleotide Mycoprotein Meal in Uric Acid Concentrations and Other Markers of Health
Brief Title: High Nucleotide Meal Consumption in Uric Acid and Metabolic Health
Acronym: TIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 170712/A/01
Record Dates: First submitted 2018-05-31; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low nucleotide meal (Placebo Comparator): Mixed meal containing mycoprotein with a reduced nucleotide content (~ 2% nucleotides)
  Interventions: Other: Low nucleotide meal
- High nucleotide meal (Experimental): Mixed meal containing mycoprotein with a high nucleotide content (~ 10% nucleotides)
  Interventions: Other: High nucleotide meal

INTERVENTIONS:
Other: Low nucleotide meal — The participants will consume a mixed meal (sandwich) containing a nucleotide depleted mycoprotein product (low in nucleotides)
  Arms: Low nucleotide meal
Other: High nucleotide meal — The participants will consume a mixed meal (sandwich) containing a non nucleotide depleted mycoprotein product (high in nucleotides)
  Arms: High nucleotide meal

SUMMARY:
The production of protein rich animal products is associated with a large environmental burden, and with ethical considerations. Additionally, the over-consumption of meat might be associated with detrimental effects to health.

Using mycoprotein, a food ingredient derived from the fermentation of a fungus, as a meat substitute could result in environmental benefits, and could have a role in managing obesity, diabetes and improving metabolic health. However, naturally produced mycoprotein has a high nucleotide content and little is known about the impact of nucleotides in uric acid levels and other health markers.

The aim of this study is to investigate the effect of a meal based on nucleotide rich mycoprotein on uric acid concentrations and other markers of health.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18 and 30

Exclusion Criteria:

* On medication (except contraception)
* Smokers
* Diagnosed with any metabolic or cardiovascular conditions
* BMI < 18 or > 30

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2018-03-14 (Actual)

PRIMARY OUTCOMES:
Changes in serum uric acid concentrations over a 24 h period | Baseline; 15, 30, 45, 60, 90, 120, 150, 180, 210 and 240 minutes after meal; 8, 12 and 24 hours after meal

SECONDARY OUTCOMES:
Blood glucose | Baseline; 15, 30, 45, 60, 90, 120, 150, 180, 210 and 240 minutes after meal; 24 hours after meal
Serum insulin | Baseline; 15, 30, 45, 60, 90, 120, 150, 180, 210 and 240 minutes after meal
Branched chained amino-acids | Baseline; 15, 30, 45, 60, 90, 120, 150, 180, 210 and 240 minutes after meal

CONTACTS AND LOCATIONS:
Locations (1):
- St Luke's Campus - University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No